CLINICAL TRIAL: NCT03244787
Title: Patient Navigation for Colorectal Cancer Screening for Patients With Mental Illness and/or Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carolina Abuelo, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016P001322
Record Dates: First submitted 2017-03-21; First posted 2017-08-10 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: ColoRectal Cancer Screening
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient navigation (Experimental): PN will contact patients during their visits to health cancer or over the phone. During this initial contact, the PN will educate patients about CRC, screening and explore their barriers to screening. The PN will coordinate scheduling of CRC screening and remind patients about the tests. PN will explain preparation for colonoscopy and whenever feasible, accompany patient to obtain the test. Further interventions may include: reminding the patient about the test, helping with translation, insurance issues, transportation, and overcoming any other system barriers as needed.
  Interventions: Behavioral: patient navigation
- usual care (No Intervention): patients randomly assigned to the control will receive usual care and be eligible for navigation after the study period.

INTERVENTIONS:
Behavioral: patient navigation — Current standard of care is for PNs to work with patients from health centers who are referred by providers. Intervention patients will appear on a PN list without any referral by providers. Control high risk patients will proceed normally and will be eligible to transfer to a PN list after the 6-month study period.
  Arms: patient navigation

SUMMARY:
The investigators propose to develop, implement, and evaluate a novel Colorectal (CRC) screening patient navigator program for patients with Mental Health (MH) and /or Substance Use Disorder (SUD) receiving care at Massachusetts General Hospital Charlestown. The study will involve randomly assigning eligible patients to early intervention or usual care/delayed intervention groups. The investigators believe this random assignment is ethical because Patient Navigation (PN) is an extremely limited resource, and all patients identified as eligible could not be contacted by the navigators in a short period of time. Thus the investigators will randomly assign access to PN during the study period, and then allow all patients to be navigated and screened after the study period is over. As a result, all eligible patients will be referred for PN, but the timing of the referral will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 50-75 years who are not up to date on CRC screening (did not have had CRCs colonoscopy in the last 10 years or sigmoidoscopy in the last 5 years or fecal occult blood within last 12 months)
* receive care at MGH Charlestown
* have documented history of MH or SUD in electronic medical record

Exclusion Criteria:

* subsequently identified as having died prior to study intervention
* patients with total colectomy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in intervention and control groups who completed any colorectal cancer screening during the six-month study period | 6 months
  To obtain the data about colorectal cancer screening we will use billing data from our institution repository. Additionally, and when/if the data is not available (percentage of colonoscopy results) we will perform EMR reviewed of trial participants.
Percentage of patients in intervention and control groups who completed any colorectal cancer screening during the six-month study period | 6 months
  To obtain the data about colorectal cancer screening we will use billing data from our institution repository. Additionally, and when/if the data is not available (percentage of fecal occult blood test results) we will perform EMR reviewed of trial participants.

SECONDARY OUTCOMES:
As-treated primary outcomes among intervention patients contacted by patient navigator. | 1 year
  Percentage of patients in intervention and control groups who completed colorectal cancer cancer screening stratified by Mental health vs Substance use disorder, language spoken, race and age (<> 65 years) during the study period
Number of cancers (stage) found in the intervention and control group during the study period | 1 year
Number of polys found in intervention polyps (histology) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Percac Lima, MD, Principal Investigator — MGH

IPD SHARING:
Plan to Share IPD: No